CLINICAL TRIAL: NCT07382674
Title: Zesty Exercise System for Therapeutic Engagement
Acronym: ZEST-E
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Georgia Clinical & Translational Science Alliance (Unknown)
Responsible Party: Principal Investigator, Madeleine Eve Hackney, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024P006965
Record Dates: First submitted 2026-01-27; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
Keywords: Exercise; Robotics; Parkinson's disease; Caregivers; Artificial Intelligence; Strength
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-Person Monitored ZEST-E Exercise (Experimental): Participants complete ZEST-E exercise sessions with a researcher or physical therapist present in the same room to provide safety oversight. All participants begin with seated exercises in week 1 and may progress to standing exercises in weeks 2 and 3 after completing a safety tutorial and demonstrating understanding of standing-exercise precautions. The researcher monitors the robot, provides instructions, and may stop the robot at any time using the run-stop button if needed.
  Interventions: Other: ZEST-E Robot-Assisted Exercise Program
- Remotely Monitored ZEST-E Exercise (Experimental): Participants complete ZEST-E exercise sessions while the researcher or physical therapist monitors the session remotely via camera from outside the room. A trained caregiver is present in the room to provide safety oversight and to activate the robot's run-stop button if needed. Participants follow the same progression from seated to standing exercises as in the in-person arm, contingent on completion of the safety tutorial and demonstration of safe technique.
  Interventions: Other: ZEST-E Robot-Assisted Exercise Program

INTERVENTIONS:
Other: ZEST-E Robot-Assisted Exercise Program — Participants complete robot-guided exercises using the ZEST-E system. Sessions include reaching, stretching, and dual-task movements for upper and lower limbs. Before each exercise, participants view a video demonstration or receive instruction from staff. ZEST-E presents targets to tap with hands, feet, or knees and uses calibration and practice trials to set positions. The robot operates with force-limited controls, back-drivable joints, and an emergency run-stop button. Participants may request to stop the robot at any time. All participants begin with seated exercises in week 1 and may progress to standing exercises in weeks 2-3 after completing a safety tutorial. Safety supports such as mats, chairs, and gait belts are used during standing tasks.
  Training will consist of 1-hour bouts, 3 times/week for 3 weeks

SUMMARY:
This study will evaluate exercise delivered through the Zesty Exercise System for Therapeutic Engagement (ZEST-E) for people with Parkinson's disease when sessions are monitored either in person or remotely. Participants will complete robot-guided exercise three times per week for three weeks. The study will assess feasibility, retention, safety, acceptability, and tolerability of remotely monitored ZEST-E and will measure changes in functional performance using the Standing Forward Reach test and the 30-Second Chair Stand test. These outcomes reflect range of motion and lower-body strength targeted by the exercise program.

DETAILED DESCRIPTION:
Parkinson's disease is associated with reduced range of motion, impaired postural control, and decreased lower-body strength, which contribute to mobility limitations and reduced functional independence. Exercise is an essential component of symptom management and has been shown to improve strength, balance, and overall physical function. Many individuals with Parkinson's disease, however, face barriers to accessing supervised exercise, including transportation challenges, limited availability of trained providers, and difficulty maintaining consistent participation. Remote delivery of structured exercise may increase accessibility, but its feasibility and safety for use with robotic exercise systems have not been fully evaluated.

The Zesty Exercise System for Therapeutic Engagement (ZEST-E) is a robotic platform designed to guide users through structured physical activity tasks that target range of motion and lower-body strength. The system provides interactive movement prompts and real-time feedback through a robotic interface. Previous work has shown that ZEST-E can be used safely and effectively in supervised settings. The current study will evaluate the use of ZEST-E when exercise sessions are monitored either in person or remotely.

Participants will complete exercise sessions three times per week for three weeks. Each session will include robot-guided movements such as forward reaching, leaning, and repeated sit-to-stand transitions. Remote monitoring will be conducted through real-time audiovisual supervision, while in-person monitoring will occur on-site. Caregivers of participants can co-enroll and will receive fall prevention training, which they will practice during the exercise sessions. Throughout the study, information will be collected on session completion, participant experience, caregiver stress, and any safety concerns.

The study will also measure changes in functional performance. The Standing Forward Reach test will be used to assess range of motion, and the 30-Second Chair Stand test will be used to assess lower-body strength. These outcomes were selected because they reflect motor abilities targeted by the ZEST-E exercise protocol. The results will provide information about the feasibility, acceptability, and safety of remotely monitored robotic exercise and will support planning for future research using this technology.

ELIGIBILITY:
Inclusion Criteria:

-Older adults with mild to moderate PD.

Exclusion Criteria:

* Acute medical illness requiring hospitalization;
* Under 40 years old;
* Uncontrolled congestive heart failure;
* History of stroke in the past three years;
* Inability to perform study procedures;
* Medical or physical conditions that would preclude participation (e.g., severe arthritis or mobility problems, uncontrolled hypertension or diabetes, renal failure, history of angina with activity);
* On medications that could adversely affect cognition, e.g.: antipsychotics, opioids, stimulants, chemotherapy;
* Psychotic disorders;
* Confounding neurologic conditions (e.g., active central nervous system opportunistic infections, seizure disorders, head injury with loss of consciousness >30 minutes, intracranial neoplasms, stroke with neurological or neuropsychiatric sequelae);
* Substance Use Disorder, Major Depressive and Generalized Anxiety Disorders within six months of evaluation;
* Hohn & Yahr > 3
* MoCA <17

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Standing Forward Reach (SFR) Test | Baseline, after 3 weeks
  This test measures forward reach distance while standing to assess range of motion and postural control. Greater reach distance indicates improved mobility.
30-Second Chair Stand Test | Baseline, after 3 weeks
  Number of full sit-to-stand repetitions completed in 30 seconds. Higher counts indicate greater lower-body strength

SECONDARY OUTCOMES:
Feasibility (Session Adherence) | Throughout 3-week intervention
  Proportion of scheduled ZEST-E sessions completed.
Retention | Throughout 3-week intervention
  Percentage of participants who complete all study assessments.
Safety (Adverse Events) | Throughout 3-week intervention
  Number and type of adverse events reported during ZEST-E sessions.
Acceptability and Tolerability | Throughout 3-week intervention
  Participant ratings of comfort, ease of use, and overall experience using standardized questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine Hackney, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, 57 Executive Park S NE, Ste 200, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No